CLINICAL TRIAL: NCT06410599
Title: Pharmacologic Treatment Augmentation in Chronic Depression "Randomized, Controlled, Double Blinded, Phase II Study"
Brief Title: Pharmacologic Treatment Augmentation in Chronic Depression
Acronym: Ket+CBASP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Center for Mental Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 519/2019AMG1; 2019-001692-37 (EudraCT Number)
Record Dates: First submitted 2024-03-05; First posted 2024-05-13 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder
Keywords: Ketamine; CBASP; Augmentation; Combination therapy; Chronic depression; MDD
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ketamine+TAU (Experimental): Combination of ketamine hydrochloride (Ketamin Inresa 2 ml) and TAU during week 4 to 6.
  TAU (treatment as usual): standard ward psychotherapeutic program (group and single sessions) with cognitive behavioural, sociotherapeutic, occupational therapy and physiotherapeutic elements.
  Interventions: Drug: Ketamine; Behavioral: TAU
- Placebo+CBASP (Placebo Comparator): Combination of placebo and CBASP during week 4 to 6.
  CBASP: In addition to standard ward psychotherapeutic program (group and single sessions) with cognitive behavioural, sociotherapeutic, occupational therapy and physiotherapeutic elements, patients in the CBASP conditions receive one CBASP group session (50 min) per week for 12 weeks. The single sessions (one 50 min and one 25 min per week) contents are CBASP-specific.
  Interventions: Drug: Placebo; Behavioral: CBASP
- Ketamine+CBASP (Experimental): Combination of ketamine hydrochloride (Ketamin Inresa 2 ml) and CBASP during week 4 to 6.
  CBASP: In addition to standard ward psychotherapeutic program (group and single sessions) with cognitive behavioural, sociotherapeutic, occupational therapy and physiotherapeutic elements, patients in the CBASP conditions receive one CBASP group session (50 min) per week for 12 weeks. The single sessions (one 50 min and one 25 min per week) contents are CBASP-specific.
  Interventions: Drug: Ketamine; Behavioral: CBASP

INTERVENTIONS:
Drug: Ketamine — Two ketamine hydrochloride (Ketamin Inresa 2 ml) infusions (interval 2-3 days) per week for three weeks, 6 infusions in total. Ketamine hydrochloride (Ketamin Inresa 2 ml) is applied continuously over a time span of 40 minutes with a subanesthetic dosage of 0.5 mg per kg body weight.
  Other Names: Ketamine hydrochloride (Ketamin Inresa 2 ml)
  Arms: Ketamine+CBASP; Ketamine+TAU
Drug: Placebo — Two times placebo (Isotone E NaCL 0.9 %) infusions (interval 2-3 days) per week for three weeks, 6 infusions in total. Placebo is applied continuously over a time span of 40 minutes.
  Other Names: Saline solution: Fresenius Kabi Deutschland GmbH Isotone E NaCL 0.9 %
  Arms: Placebo+CBASP
Behavioral: CBASP — In addition to standard ward psychotherapeutic program (group and single sessions) with cognitive behavioural, sociotherapeutic, occupational therapy and physiotherapeutic elements, patients in the CBASP conditions receive one CBASP group session (50 min) per week for 12 weeks. The single sessions (one 50 min and one 25 min per week) contents are CBASP-specific.
  Other Names: Cognitive Behavioral Analysis System of Psychotherapy
  Arms: Ketamine+CBASP; Placebo+CBASP
Behavioral: TAU — Standard ward psychotherapeutic program (group and single sessions) with cognitive behavioural, sociotherapeutic, occupational therapy and physiotherapeutic elements.
  Other Names: Treatment as usual
  Arms: Ketamine+TAU

SUMMARY:
To enroll in this clinical trial, prospective participants must meet stringent criteria. The participants need to fall within the age range of 18 to 64 and exhibit chronic depression at therapy resistance stage 2. This stage signifies that the participants have undergone unsuccessful treatment with at least two different antidepressants, despite adequate dosage and duration. Moreover, the participants should have engaged in at least 12 sessions of psychotherapy without experiencing significant relief from depressive symptoms. Additionally, participants must demonstrate the cognitive capacity to provide informed consent.

Upon expressing interest in the study and consenting to participate, individuals undergo a thorough screening process. This screening encompasses a comprehensive clinical interview to assess medical and psychiatric history, as well as various medical tests. These tests include physical examinations, blood draws (which may include pregnancy tests for female participants), and electrocardiograms (ECGs) to evaluate heart function. Following the screening, participants are randomly assigned to one of three different treatment groups (Ketamine +TAU; Ketamine+CBASP, Placebo+CBASP).

The study protocol involves a combination of psychotherapeutic treatment and either ketamine infusions or placebo. Throughout the study period, participants are subject to regular data collection, including psychological assessments, blood samples, and magnetic resonance imaging (MRI) scans. Participants' responses to treatment, as well as any changes in symptoms or side effects, are closely monitored.

After completing the study, participants are offered follow-up therapy as part of standard care. MRI scans are conducted to examine changes in brain activity associated with treatment response and depressive symptomatology, particularly focusing on alterations in neural circuitry and thought processes. Additionally, participants are encouraged to report any changes in medication regimen or other treatments received during the study period.

DETAILED DESCRIPTION:
To participate in this clinical trial, one must have reached the age of 18 at the time of enrollment and not have exceeded the age of 64. Additionally, the pilot study is designed for patients with chronic depression who are in therapy resistance stage 2. Therapy resistance stage 2 means that one has taken at least 2 antidepressants from two different classes in sufficient dosage over a sufficient period of time without experiencing significant and sustainable improvement in depressive symptoms. Furthermore, one should have received at least 12 sessions of psychotherapy (psychoanalysis, psychodynamic psychotherapy, or cognitive behavioral therapy) without significant and sustainable improvement in depressive symptoms. Also, one must have the capacity to consent.

Those interested in participating in this study must have provided written consent to participate. A screening takes place to check the criteria for study participation using a clinical interview. The clinical interview collects information about current and previous physical and mental symptoms or diagnoses and treatments and lasts approximately 100 minutes. Additionally, a physical examination, a blood draw of approximately 20 ml, and an electrocardiogram (ECG) to determine heart activity are performed.

If one meets the inclusion criteria and no exclusion criteria are present, one can participate in the study and will be randomly assigned to one of the three treatment groups (Ketamine+TAU; Ketamine+CBASP, Placebo+CBASP). Participants are being told what type of psychotherapy the participant will receive. If one is assigned to one of the CBASP groups, neither the participant nor the treatment team will be informed whether the participant is receiving ketamine or placebo.

Once the group assignment is made, further data is collected in the first study week. In week 2, the psychotherapeutic treatment begins with a two-week introductory phase. Psychotherapy includes two individual sessions per week as well as group therapies. At the end of the introductory phase, further data collection takes place.

In week 3, additional data is collected, and a blood draw is performed to repeat the pregnancy test. Subsequently (weeks 4-6), one is treated with an infusion twice a week for three weeks (ketamine or placebo). The infusions within a week are spaced 2-3 days apart and each lasts approximately 40 minutes. Psychotherapy continues during these three weeks. After completing the combination treatment of study medication/placebo and psychotherapy, further data is collected, and psychotherapy continues for another 6 weeks (weeks 7-12). After that, the treatment as part of the study is completed.

To optimize treatment success and prevent relapses, an appropriate follow-up therapy is planned and initiated in consultation with the study therapist, depending on the individual development during the study therapy. Three months after completing the study therapy, the final data collection is carried out. Throughout the entire study, a total of 9 blood draws are performed.

Psychotherapy, administration of study medication/placebo, and data collection are carried out at the study site. Existing medication may continue to be taken during the study and will be optimized as needed. If medication with benzodiazepines is prescribed, it cannot be taken on the day before the infusion or on the day of the infusion.

The first blood draw and urine sample are used to get an impression of one's overall health status and thus assess whether participation in the study is possible or permissible according to the inclusion and exclusion criteria. In addition, a drug screening is performed on the urine sample to exclude acute substance abuse (alcohol, drugs), and a pregnancy test is performed based on the blood sample.

In the event of discontinuation of the study, follow-up treatment will be offered within the standard therapy for depressive disorders.

Additional medications (including over-the-counter ones) of which the investigator is not yet aware may only be taken in emergencies after consulting the investigator. If one is being treated by other doctors, the other doctors must be informed about participation in the clinical trial. The investigator must also be informed about any medical treatment received from another doctor during the clinical trial. One will receive a study ID card, which should always be carried for emergencies.

The fMRI examination in weeks 3 and 12 is performed to assess changes in brain activity during treatment and in relation to changes in depressive symptoms. Additionally, the relationship between mind wandering and brain activity in the presence of depressive illness is analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 64 years at the time of study inclusion.
* Diagnosis of chronic depression: recurrent depressive disorder, severe or moderate episodes (no full remission between the episodes according to DSM-IV-TR (Falkai et al., 2015) [no distinct depressive symptoms for at least two months]) or acute depressive episode lasting two or more years
* Treatment resistance stage 2 according to (Thase and Rush, 1997): Patient's symptoms fulfil the criteria of chronic depression listed above even after at least two appropriate treatment attempts with two antidepressant medicaments from two different effect categories
* Patient's symptoms fulfil the criteria of chronic depression listed above even after executing at least 12 sessions of psychotherapeutic treatment (psychoanalysis, depth psychology-based psychotherapy or cognitive behaviour therapy)
* Understand and voluntarily sign an informed consent document prior to any study related assessments/ procedures.
* Able to adhere to the study visit schedule and other protocol requirements.
* Females of childbearing potential (FCBP) must agree to utilize two reliable forms of contraception simultaneously or practice complete abstinence from heterosexual contact from study start until 28 days after the last infusion.
* Males must agree to use a latex condom during any sexual contact with FCBP from the first infusion until 65 days after the last infusion, even if the person has undergone a successful vasectomy to refrain from donating semen or sperm from the first infusion until 65 days after the last infusion.
* All subjects must agree to refrain from donating blood from the first infusion until 28 days after last infusion.
* All subjects must agree not to share medication.

Exclusion Criteria:

* Acute substance misuse as primary diagnosis (assessed by the Structured Clinical Interview for DSM-V (SKID, Wittchen et al., 1997))
* Neurologic disorders: Stroke, cerebral ischemia, tumor, cerebral infection, autoimmune disease (according to clinical interview)
* Disorders with increase of intracranial pressure, e. g. due to head injury (according to clinical interview)
* Circulatory disturbance in the brain (according to clinical interview)
* Pregnant or lactating females
* Participation in any clinical study or having taken any investigational therapy, which would interfere with the study's primary end point
* Epilepsy (according to clinical interview)
* History of hypersensitivity to an investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product (according to clinical interview)
* Pre-treatment with ketamine hydrochloride (Ketamin Inresa 2 ml) and/ or - CBASP (according to clinical interview)
* Not or insufficiently treated hypertonia (subject will be excluded if repeated measures (3 times/ day) show values greater than 150 mmHg systolic or 100 mmHg diastolic blood pressure or if a lifetime diagnosis of hypertonia is reported)
* Not or insufficiently treated hyperthyroidism (according to clinical interview)
* Heartache due to insufficient blood circulation (unstable angina pectoris) or heart muscle infarct (myocardia infarct) during the last six months (according to clinical interview)
* Increased intraocular pressure (glaucoma) and perforating eye injury (according to clinical interview)
* Interventions in the area of the upper respiratory passages (according to clinical interview)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change of depressive symptoms assessed with Montgomery-Åsberg Depression Rating Scale (MADRS) between start and end of treatment in a group comparison | 3 months after enrollment
  Change of depressive symptoms (assessed with Montgomery-Åsberg Depression Rating Scale (MADRS), Schmidtke et al., 1988) between start of and six weeks after end of combination treatment (Δ t1-t3) in group 1 (ketamine plus CBASP) vs. group 2 (placebo plus CBASP) and in group 1 vs. group 3 (ketamine plus TAU). Lower scores indicate better treatment outcome.

SECONDARY OUTCOMES:
Change of depressive symptoms assessed with Montgomery-Åsberg Depression Rating Scale (MADRS) in a group comparison | 6 months after enrollment
  Change of depressive Symptoms (assessed with Montgomery-Åsberg Depression Rating Scale (MADRS), Schmidtke et al., 1988) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up). Lower scores indicate better treatment outcome.
Change of depressive symptoms of self-reported depressive symptoms (assessed with Beck-Depression-Inventory (BDI) in a group comparison | 3 months after enrollment
  Change of self-reported depressive symptoms assessed with Beck-Depression-Inventory (BDI), Beck et al., 2001) between start of and six weeks after end of combination treatment (Δ t1-t3) in group 1 (ketamine plus CBASP) vs. group 2 (placebo plus CBASP) and in group 1 vs. group 3 (ketamine plus treatment as usual (TAU). Lower scores indicate better treatment outcome.

OTHER OUTCOMES:
Pearson/Spearman correlation between actual number of single and group sessions and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between actual number of single and group sessions and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between actual session contents and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between actual session contents and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between training level and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between training level and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between antidepressant medication (screening log) and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between antidepressant medication (screening log) and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between psychosocial support FSozU (Fragebogen zur Sozialen Unterstützung, Fydrich et al., 1999) and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between psychosocial support FSozU (Fragebogen zur Sozialen Unterstützung, Fydrich et al., 1999) and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between psychosocial functioning (Global Assessment of Functioning, Monrad Aas, 2014)) and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between psychosocial functioning (Global Assessment of Functioning, Monrad Aas, 2014)) and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between severity of depression (MADRS) and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between severity of depression (MADRS) and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between depressive subtype (MADRS) and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between depressive subtype (MADRS) and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between comorbid disorders (SKID) and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between comorbid disorders (SKID) and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between quality of therapeutic alliance and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between quality of therapeutic alliance and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between premorbid intelligence (MWT-B (Mehrfachwahl- Wortschatz-Intelligenztest, Lehrl, 2005)) and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between premorbid intelligence (MWT-B (Mehrfachwahl- Wortschatz-Intelligenztest, Lehrl, 2005)) and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between childhood traumatization (CTQ (Childhood Trauma Questionnaire, Wingenfeld et al., 2010)) and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between childhood traumatization (CTQ (Childhood Trauma Questionnaire, Wingenfeld et al., 2010)) and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between Brain Derived Neurotrophic Factor (BDNF) concentration and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between Brain Derived Neurotrophic Factor (BDNF) concentration and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between brain activity (resting-state fMRI) and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between brain activity (resting-state fMRI) and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between quality of life (World Health Organization WHOQOL-BREF quality of life assessment, WHO, 1998) and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between quality of life (World Health Organization WHOQOL-BREF quality of life assessment, WHO, 1998) and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between self-esteem (State self-esteem scale, Heatherton and Polivy, 1991) and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between self-esteem (State self-esteem scale, Heatherton and Polivy, 1991) and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between emotional regulation (Heidelberger Form for Emotion Regulation Strategies (H-FERST), Izadpanah et al., 2019) and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between emotional regulation (Heidelberger Form for Emotion Regulation Strategies (H-FERST), Izadpanah et al., 2019) and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between emotional regulation (emotional regulation fMRI paradigm) and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between emotional regulation (emotional regulation fMRI paradigm) and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between emotional state (PANAS, Watson et al., 1988) and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between emotional state (PANAS, Watson et al., 1988) and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.
Pearson/Spearman correlation between emotional state Emotional Self Rating (ESR, Schneider et al., 1995) and changes in depressive symptoms (as assessed by MADRS) in the different treatment groups. | 6 months after enrollment
  Pearson/Spearman correlation between emotional state Emotional Self Rating (ESR, Schneider et al., 1995) and changes (delta between timepoints) in depressive symptoms (as assessed by MADRS) between start of combination treatment and three months after the end of study treatment (Δ t1- follow up) in the different treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Walter, Prof. Dr., Principal Investigator — Universitätsklinikum Jena - Klinik für Psychiatrie und Psychotherapie; Andreas J Fallgatter, Prof. Dr., Principal Investigator — Universitätsklinikum Tübingen - Klinik für Psychiatrie und Psychotherapie
Locations (2):
- Germany (2):
  - Universitätsklinikum Tübingen - Klinik für Psychiatrie und Psychotherapie, Tübingen, Baden-Würtemberg
  - Universitätsklinikum Jena - Klinik für Psychiatrie und Psychotherapie, Jena, Thuringia

IPD SHARING:
Plan to Share IPD: No